CLINICAL TRIAL: NCT03917628
Title: Pharmacokinetics and Safety of SCT630 in Healthy Subjects: a Randomized, Double-blind, Single Dose Clinical Phase I Study.
Brief Title: Pharmacokinetics and Safety in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT630PS01
Record Dates: First submitted 2019-04-14; First posted 2019-04-17 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT630 (Experimental): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing SCT630
  Interventions: Drug: SCT630
- adalimumab-EU source (Active Comparator): Subject to receive one subcutaneous (s.c.) injection from a prefilled syringe containing adalimumab-EU source
  Interventions: Drug: adalimumab-EU source

INTERVENTIONS:
Drug: SCT630 — SCT630 single s.c. injection
  Arms: SCT630
Drug: adalimumab-EU source — adalimumab-EU source single s.c. injection
  Arms: adalimumab-EU source

SUMMARY:
Investigate the pharmacokinetics, safety and tolerability of SCT630 and to establish pharmacokinetic similarity of SCT630 to adalimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged 18 to 45 years
2. Body mass index (BMI) between 19 and 26 kg/m2
3. Normal or clinically acceptable physical examination, clinical laboratory values, ECG, chest X-ray and vital signs at screening and baseline.
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

1. History or evidence of a clinically significant disorder, condition, or disease that would have posed a risk to subject safety or would have interfered with the study evaluation, procedures, or study completion in the opinion of the investigator.
2. Evidence of any bacterial, viral, parasitic, systemic fungal infections, or infections due to other opportunistic pathogens within the 30 days prior to investigational product administration.
3. History of tuberculosis,positive test for Interferon-gamma-release assay,or suffering from active tuberculosis or latent tuberculosis infection.
4. History of malignancy of any type, other than surgically excised nonmelanomatous skin cancers, within 5 years prior to investigational product administration.
5. Positive test for HIV antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies at screening.
6. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients).
7. Quantification of Hepatitis B virus DNA is greater than the upper limit of normal value.
8. Received biologics or live vaccines ≤3 months prior to investigational product administration.
9. Intake of an investigational drug in another trial within three months prior to investigational product administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
AUC0-tz | at -1 hour (h) (pre dosing) and 8, 24, 48, 72, 96, 120, 144, 168, 192, 336, 504, 672, 840, 1008,1344 h post dosing and on day 71 post dosing.
  Area Under the Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC0-tz) of SCT630 and EU-licensed Humira
Cmax | at -1 hour (h) (pre dosing) and 8, 24, 48, 72, 96, 120, 144, 168, 192, 336, 504, 672, 840, 1008,1344 h post dosing and on day 71 post dosing.
  Maximum Concentration (Cmax) of SCT630 and EU-licensed Humira

SECONDARY OUTCOMES:
AUC 0-∞ | at -1 hour (h) (pre dosing) and 8, 24, 48, 72, 96, 120, 144, 168, 192, 336, 504, 672, 840, 1008,1344 h post dosing and on day 71 post dosing.
  Area Under the Concentration Time Curve (AUC) From Time Zero to Infinity (AUC 0-∞) of SCT630 and EU-licensed Humira
Tmax | at -1 hour (h) (pre dosing) and 8, 24, 48, 72, 96, 120, 144, 168, 192, 336, 504, 672, 840, 1008,1344 h post dosing and on day 71 post dosing.
  Time to the Maximum Concentration of SCT630 and EU-licensed Humira
t1/2 | at -1 hour (h) (pre dosing) and 8, 24, 48, 72, 96, 120, 144, 168, 192, 336, 504, 672, 840, 1008,1344 h post dosing and on day 71 post dosing.
  Elimination Phase Half-life of SCT630 and EU-licensed Humira
λz | Day 1 through Day 71
  λz of SCT630 and EU-licensed Humira
CL | Day 1 through Day 71
  Clearance rate of the SCT630 and EU-licensed Humira
Vd | Day 1 through Day 71
  Apparent volume of distribution (Vd) of the SCT630 and EU-licensed Humira
Number (Proportion) of Subjects With Drug Related Adverse Events | Day 1 through Day 71
Positive rate of ADA and NAb | Day 1 through Day 71
  Comparision of the positive rate of ADA and NAb between the SCT630 and EU-licensed Humira

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing SHIJITAN Hospital, Beijing, Beijing Municipality, China